CLINICAL TRIAL: NCT07106983
Title: Gagging and Feelings of Disgust: Forgotten Reactions in Dental Treatment?
Status: Completed | Type: Observational
Sponsor: Oral Health Centre of Expertise in Western Norway (Other)
Responsible Party: Sponsor
Other Study IDs: 458062
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2022-09

CONDITIONS: Gagging; Disgust
Keywords: gagging; disgust; dental anxiety; abuse
MeSH Terms: conditions — Gagging | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention (observational study) — Observational survey only

SUMMARY:
This cross-sectional study aims to validate two questionnaires: one measuring gagging related to dental treatment, and another assessing feelings of disgust and aversion. It also explores associations with self-reported experiences, including dental fear and a history of abuse.

Gagging and disgust in dental settings are complex reactions that may hinder access to necessary care, affecting oral health and quality of life.

The study includes two anonymous surveys:

* Young adults from Vestland County, recruited via SMS
* Dental and dental hygiene students at the University of Bergen

Validated instruments were used, including DPSS-R, Predictive Gagging Survey, GPA, MDAS, and IOIF-s.

DETAILED DESCRIPTION:
This study aims to validate two questionnaires: one assessing gagging related to dental treatment, and another measuring feelings of disgust and aversion in dental treatment. Additionally, the study explores associations between these responses and self-reported life experiences, including sexual abuse and dental fear.

Gagging and disgust in dental settings are complex responses with both biological and psychological components. For affected individuals, these reactions may interfere with the ability to receive necessary dental care, with potential negative consequences for oral health and quality of life.

This quantitative cross-sectional study includes data that were partially used in a master's thesis at the University of Bergen (2023), conducted as part of the broader research project. The study consists of two sub-studies:

Sub-study I: Young adults from Vestland County were recruited via SMS to complete an anonymous online survey.

Sub-study II: Dental and dental hygiene students at the University of Bergen were invited via the learning platform Mitt UiB.

The surveys collected data on participants' experiences with gagging, dental fear, fear of intraoral injections, and disgust/aversion. Psychometric instruments used included the Disgust Propensity and Sensitivity - Revised (DPSS-R), The Predictive Gagging Survey, Gagging Problem Assessment (GPA), Modified Dental Anxiety Scale (MDAS), and Intra- Oral Injection Fear scale (IOIF).

The study contributes to the validation of tools for assessing gagging and disgust in dental care, and increases knowledge about possible associations between gagging, aversion, dental anxiety, and history of abuse.

ELIGIBILITY:
* Young adults born between 2000 and 2001, recruited from the Public Dental Health Service in Vestland County
* All dental and dental hygienist students at the University of Bergen in 2022

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * Young adults born between 2000 and 2001, recruited from the Public Dental Health Service in Vestland County
  * All dental and dental hygienist students at the University of Bergen in 2022
Sampling Method: Non-Probability Sample
Enrollment: 1472 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
Validation of a Questionnaire Assessing Gag Reflex During Dental Treatment | From data collection start in October 2022 until the end of data collection December 2022.
  Evaluation of the questionnaire's validity in measuring the prevalence of gagging during dental procedures in young adults in Western Norway.
Validation of a Questionnaire Assessing Disgust During Dental Treatment | From data collection start in October 2022 until the end of data collection December 2022.
  Evaluation of the questionnaire's validity in measuring the prevalence of disgust response during dental procedures in young adults in Western Norway.
The prevalence of gagging | From data collection start in October 2022 until the end of data collection December 2022.
  Assessing the prevalence of gagging in young adults in Westen Norway.
The prevalence of disgust | From data collection start in October 2022 until the end of data collection December 2022.
  Assessing the prevalence of disgust among young adults in Western Norway

SECONDARY OUTCOMES:
Association Between Gag Reflex and Self-Reported Life Experiences | From data collection start in October 2022 until the end of data collection December 2022.
  Examination of the correlation between self-reported instances of gagging during dental treatment and past life experiences, such as sexual abuse and dental anxiety.
Prevalence of Gag Reflex and feelings of disgust Among Dental and Dental Hygiene Students | From data collection start in October 2022 until the end of data collection December 2022.
  Measurement of the prevalence of gagging and disgust responses during dental treatment among dental and dental hygienist students at the University of Bergen.

CONTACTS AND LOCATIONS:
Locations (1):
- The Oral Health Centre of Expertise in Western Norway, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No
Individual participant data from this study will not be shared due to privacy concerns and in accordance with applicable laws and regulations.